CLINICAL TRIAL: NCT07143838
Title: Investigating Slow Wave Sleep Enhancement to Improve Cognitive Function in Adults With Depression
Brief Title: Enhancing Slow Wave Sleep in Depression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00134801
Record Dates: First submitted 2025-08-18; First posted 2025-08-27 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-07

CONDITIONS: Depression - Major Depressive Disorder
Keywords: Sleep; Depression
MeSH Terms: conditions — Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Transcranial Electrical Stimulation (TES) (Experimental): All participants will receive transcranial electrical stimulation (TES) during sleep
  Interventions: Device: Transcranial Electrical Stimulation (TES)

INTERVENTIONS:
Device: Transcranial Electrical Stimulation (TES) — Using the Sleep WISP device, transcranial electrical stimulation will be delivered during sleep as 0.5 Hz sine wave, 0.5 mA, between frontal (frontopolar and inferior lateral frontal) and posterior (mastoid and occipital) electrodes.
  Other Names: Sleep WISP (Wireless Interface Sensor Pod)

SUMMARY:
The goal of this pilot study is to determine if non-invasive brain stimulation during sleep can increase deep sleep in adults with depression. It will also determine if increased deep sleep improves cognitive performance and mood ratings. Participants will be asked to wear a non-invasive device that records their brain activity and delivers transcranial electrical stimulation during sleep. Participants will also wear an actigraphy watch that measures activity levels throughout the study. In addition, participants will complete several cognitive assessments and mood and sleep questionnaires throughout the study.

DETAILED DESCRIPTION:
The purpose of this pilot study is to determine if non-invasive transcranial electrical stimulation (TES) delivered during slow-wave sleep (SWS) can enhance this stage of sleep in people with depression. Individuals with depression frequently report sleep and cognitive disturbances as symptoms associated with their depression. However, common anti-depressants often fail to improve these symptoms. A pilot study with this device showed that TES can enhance slow wave sleep in healthy individuals. This study aims to evaluate if TES will enhance deep sleep in individuals with depression as well, leading to improved sleep outcomes and potentially improving cognitive performance and mood symptoms.

This study proposes to conduct using the Sleep WISP device (Brain Electrophysiology Laboratory (BEL), Eugene, OR). Using this non-invasive device, the study will record brain activity using a technique called electroencephalography (EEG) that will be automatically scored in real-time to determine the stage of sleep. After the participant enters stable slow wave sleep, the headband will deliver the TES current (0.5-1 milliampere (mA) total) directly to the scalp through pre-set electrodes. The stimulation will be applied for 5 cycles of 5 minutes of stimulation, 1 minute of no stimulation (30 minutes total). This level and location of stimulation was previously shown as sufficient to increase SWS.

After screening and enrolling in the study, participants will have up to three nights of baseline recordings using the WISP headband to ensure successful baseline measurements are recorded. Participants will then receive TES nightly for two weeks. Participants will also wear an actigraphy watch and keep a sleep diary throughout the duration of the study. Finally, participants will complete several cognitive assessments and sleep and mood questionnaires throughout the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Ability to complete overnight sleep study including placement of EEG leads
* Ability to read and understand English.
* Moderate depression
* Self-reported cognitive complaints

Exclusion Criteria:

* Previous adverse reaction to transcranial electrical stimulation
* Presence of implanted devices (e.g. intracranial device, cochlear implant)
* Presence of metal in head (e.g. surgical clip)
* Sensitivity or allergy to silver
* Presence of significant neurologic disease (e.g. Parkinson's disease, epilepsy/seizure disorder, severe migraine disorder)
* History of significant head trauma
* History of stroke or other ischemic event
* Diagnosed with schizophrenia, bipolar disorder, substance use disorder, or presence of current suicidal ideation
* Currently taking medications that could alter EEG or cognitive function
* Presence of severe insomnia
* Presence of severe, untreated sleep apnea
* Currently pregnant
* Planned travel outside time zone during the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Duration of Stage N3 Sleep | From baseline to week 3
  Change in number of minutes of stage N3 sleep across the night
Percentage of N3 Sleep | From baseline to week 3
  Change in percentage of stage N3 sleep across the night relative to total sleep time

SECONDARY OUTCOMES:
Word Pairs Memory Task | Baseline, week 2, week 3
  Participants are presented with 44 word-pairs to learn during an encoding phase and immediately tested by presenting one word and being asked to recall the paired word. Participants are tested again in the morning in the same way - one word of the pair is presented and they are asked to recall the other. To avoid recency and priming effects, the first 4 and last 4 word pairs presented are not scored. Participants are scored on accuracy (0-36 words). A smaller decline in accuracy from the immediate recall (evening) to delayed recall phase (morning) indicates better verbal memory performance.
Choice Reaction Time (CRT) | Baseline, week 2, week 3
  CRT measures the time it takes for a person to respond to a stimulus when there are multiple possible responses to choose from. It is a measure of how quickly someone can process information, make a decision, and initiate a motor response. Participants are presented with 20 trials of stimuli to respond to. The test is scored on average reaction time where a longer reaction time indicates worse processing speed performance.
Digit Symbol Substitution Test (DSST) | Baseline, week 2, week 3
  133-item neuropsychological assessment that measures cognitive functions like processing speed, attention, and visuoperceptual skills. It involves matching symbols to numbers based on a provided key and is often used to assess cognitive impairment. The number of correct symbols within 120 seconds constitutes the score (0-133 max score) where a lower score represents greater impairment in processing speed and attention.
One-Back Working Memory Test | Baseline, week 2, week 3
  Cognitive test that assesses an individual's ability to hold and manipulate information in their short-term memory. The one-back working memory test is scored by assessing both accuracy and average response time. Accuracy is measured as the percentage of correct responses (hits) to target stimuli, while response time reflects the average speed at which participants identify matches. Higher accuracy and faster response times generally indicate better working memory performance. Participants are presented with 20 total trials (potential accuracy score, 0-20; potential reaction time 0-3 seconds). Both the accuracy and reaction time scores are z-scored and then combined to create a single composite score for the test.
Trail Making Test B (TMT-B) | Baseline, week 2, week 3
  TMT-B assesses cognitive flexibility, the ability to switch between different mental sets (in this case, numbers and letters). It also evaluates visual scanning and attention. The test taker is given a sheet of paper with 25 circles, each containing a number (1-13) or a letter (A-L). They must draw a line connecting the circles in ascending order, alternating between numbers and letters (1-A-2-B, and so on). The primary score is the time it takes to complete the task (0-300 seconds). Longer duration to complete indicates greater impairment in cognitive flexibility and attention.
Perceived Deficits Questionnaire 5 (PDQ-5) | Baseline, week 2, week 3
  5-item questionnaire with total score range 0-20. Higher score indicates greater perceived deficit.
Center for Epidemiologic Studies Depression Scale (CES-D) | Baseline, week 2, week 3
  20 items with total score range 0-60. Higher scores indicate greater severity of depressive symptoms.
Patient Health Questionnaire (PHQ-9) | Baseline, week 2, week 3
  9 items with total score range 0-27. Higher scores indicate greater severity of depressive symptoms.

OTHER OUTCOMES:
Epworth Sleepiness Scale | Baseline, Week 3
  The Epworth Sleepiness Scale (ESS) is an 8-item self-administered questionnaire to assess an individual's level of daytime sleepiness. Scores range from 0 to 24, with higher scores indicating greater daytime sleepiness. A score of 10 or higher generally suggests excessive daytime sleepiness, possibly indicating a sleep disorder.
Pittsburgh Sleep Quality Index | Baseline, Week 3
  The Pittsburgh Sleep Quality Index (PSQI) is a 19-item self-report questionnaire used to assess sleep quality and disturbances over a one-month period. Scores range from 0-21, where a higher score indicates more severe sleep disturbance. Generally, a global score of greater than 5 indicates poor sleep quality.
Morningness-Eveningness Questionnaire | Baseline
  The Morningness-Eveningness Questionnaire (MEQ) is a 19-item subjective assessment designed to assess individual differences in morningness and eveningness - the degree to which respondents are active and alert at certain times of day. The MEQ is scored by summing the responses to 19 questions, with each question offering multiple choice answers that are assigned numerical values. Scores range from 16 to 86, with lower scores indicating an "evening" chronotype and higher scores indicating a "morning" chronotype.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Benca, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hathaway E, Morgan K, Carson M, Shusterman R, Fernandez-Corazza M, Luu P, Tucker DM. Transcranial Electrical Stimulation targeting limbic cortex increases the duration of human deep sleep. Sleep Med. 2021 May;81:350-357. doi: 10.1016/j.sleep.2021.03.001. Epub 2021 Mar 8. PMID 33812203
- [Background] Peterson MJ, Benca RM. Sleep in mood disorders. Psychiatr Clin North Am. 2006 Dec;29(4):1009-32; abstract ix. doi: 10.1016/j.psc.2006.09.003. PMID 17118279
- [Background] Benca RM, Obermeyer WH, Thisted RA, Gillin JC. Sleep and psychiatric disorders. A meta-analysis. Arch Gen Psychiatry. 1992 Aug;49(8):651-68; discussion 669-70. doi: 10.1001/archpsyc.1992.01820080059010. PMID 1386215